CLINICAL TRIAL: NCT04845360
Title: China Medical University, Taiwan
Brief Title: Pulse Spectrum Analysis of Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: /CMUH108-REC1-135
Record Dates: First submitted 2021-04-06; First posted 2021-04-15 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Harmonic Wave
Keywords: Pulse diagnosis; Arterial pulse; Fourier transform; Gender differences; Pregnancy; Harmonics; Gestation
MeSH Terms: interventions — Transducers, Pressure

STUDY DESIGN:
Intervention Model Description: We performed non--invasive recording of the radial arterial pulses for 36 pregnant women, and then compared the harmonics of the radial arterial pulse after Fourier transformation with those of 50 healthy nonpregnant women (controls).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pregnancy and differences in gender can be found in the radial arterial pulse (Experimental): Establishing the meridian through harmonics of blood pressure waves could be a powerful tool to qualitatively and quantitatively indicate physiologic and pathologic factors.
  Interventions: Device: pressure transducer (PSL-200GL, Kyowa Electronic Instrument Co. Ltd., Japan)

INTERVENTIONS:
Device: pressure transducer (PSL-200GL, Kyowa Electronic Instrument Co. Ltd., Japan) — The device was fixed on the patient's skin with Scotch™ tape, along with an adjustable belt with a small button to give suitable pressure on the transducer.

SUMMARY:
ABSTRACT Background: Pulse diagnosis is a core clinical technique used in Chinese medicine to establish a patient's physiologic or pathologic status.

Methods: We performed non--invasive recording of the radial arterial pulses for 36 pregnant women, and then compared the harmonics of the radial arterial pulse after Fourier transformation with those of 50 healthy nonpregnant women (controls).

DETAILED DESCRIPTION:
The importance of information within arterial pulse waves has long been recognized in clinical medicine (Mohamed, 1872). Arterial pulse wave analysis has been employed widely in clinical practice, such as in cases of hypertension, cardiac failure, and ageing (O'Rourke, et al., 2001). Our previous studies revealed that the pulse spectrum of the radial arterial pulse could be highly correlated among patients with abnormal liver function (Wang, et al., 1996, Wang, et al., 1996). In addition, the specific Fourier components in the pulse provide more physiologic information than do systolic and diastolic blood pressure measurements during the process of dying (Kuo, et al., 2004, Kuo, et al., 2005). Recently, the fourth harmonic of the radial pulse wave has been shown to predict adverse cardiac events in asymptomatic patients with type 2 diabetes (Chang, et al., 2019)and pulse spectrum analysis has facilitated the diagnosis of coronary artery disease (Huang et al., 2019) One key method in Chinese medicine is using the harmonics of the arterial pulse to provide meridian information that can then be used to reveal a patient's physiologic and pathologic condition (Wang, et al., 2010).

In the clinic, the most dramatic physiologic event is pregnancy. Many documents discuss these issues in Chinese Medicine; for example, as stated in the bible of Chinese Medicine, Huang-Ti-Nei-Ching (1981),: "Normal pulse but appears weak, pregnancy" and "Significantly moving in Shaoyin (少陰) meridian, pregnancy." "Pulse Classics" (Wang, 2000) Another example is "Differential diagnosis of the Chi (尺), in which the pulse can detect the gender of the fetus, left larger than right is male; right larger than left is female." There is much information about pregnancy in pulse diagnosis, which has been practiced in clinics for a very long time. In fact, this practice has been used so long and so often that it has become difficult to determine the exact meaning and the accuracy of other practical approaches. Pulse diagnosis is the most important work to build the practicing definition of physiology, pathology, and diagnosis in the study of Chinese medicine.

In a previous study, we found that each organ and its related meridian are in resonance with a specific Fourier component of pressure wave (Wang, et al., 1994, Wang, et al., 1991). We also ascertained that the lower-frequency components were referred to as "Yin" and the higher ones as "Yang," and figured out the scientific meaning for the failure of hepatic, renal, or splenic Chi in the pulse (Kuo, et al., 2005). The meridian information gained through measuring the harmonics of blood pressure gives us qualitative and quantitative ways to realize the abstract statement in classic Chinese medicine. In the current study, we analyzed the blood pressure (BP) pulse of pregnant women to verify the information recorded with classic methods. We hypothesized that harmonics could be physiologic indicators corresponding with the gestation process. If we could find the relationship between harmonic information and pregnancy, we could confirm that the physiologic difference comes from the meridian, and could then precisely apply this information in the clinic.

ELIGIBILITY:
Inclusion Criteria:

* pregnant patients who visited the outpatient department (OPD)

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnancy
Enrollment: 86 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
Meridian Differences in the Radial Pulse Wave in Pregnancy and with the Gender of the Fetus | two-year study
  Results showed in the right hand, the first and second harmonics were significantly higher among the pregnant group; in the left hand, the second (P < 0.01) and fourth (P < 0.05) harmonics were significantly higher among the pregnant group; 8 other harmonics were significantly lower among pregnant group (P <0.01). When we compared the synchronously recorded data from the right and left radial arterial pulses, significant differences by gender of the fetus was found for both hands. The first, second (P < 0.01), and third (P < 0.05) harmonic differences of the left and right radial arterial pulses were significantly higher when the fetus was male. The second harmonic was the most significant indicator of gender and monthly growth of the fetus.
  Noninvasive pulse pressures of the right and left radical arteries were synchronously obtained at each OPD visit with a pressure transducer (PSL-200GL, Kyowa Electronic Instrument Co. Ltd., Japan).

CONTACTS AND LOCATIONS:
Locations (1):
- Yu- Cheng Kuo, Taipei, Taiwan